CLINICAL TRIAL: NCT03981367
Title: Frequency of External Root Resorption and Distal Caries in Mandibular Second Molars Associated With Mandibular Impacted Third Molars in a Sample of Egyptian Population Using CBCT: A Hospital-Based Cross-Sectional Study
Brief Title: Frequency of External Root Resorption in Mandibular Second Molars Associated With Mandibular Impacted Third Molars Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawan Abdel Wahhab Bahaa Eldin Elkassas, Principal Investigator, Cairo University
Other Study IDs: RAD2:8:11
Record Dates: First submitted 2019-06-03; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Root Resorption; Distal Caries
Keywords: External root resorption; Distal caries; Mandibular third molar; Mandibular second molar; Cone beam computed tomography
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of external root resorption and distal caries in mandibular second molars associated with impacted mandibular third molars will be detected in addition to the association of the risk factors.

DETAILED DESCRIPTION:
Settings:

The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo, Egypt.

CBCT images will be obtained from Egyptian patients who had CBCT examination as part of their dental examination, diagnosis or treatment planning.

Variables:

1. Angulation of the third molar according to Winter's classification (vertical/mesio-angular/disto-angular/horizontal).
2. Position of impacted mandibular third molar according to Pell and Gregory21 classification. (Position A, position B, position C)
3. Age.
4. Gender.

3. Data Sources / Measurements:

* Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.
* All the CBCT examinations will be scanned using CBCT Software (Planmeca Romexis Viewer).
* CBCT images will be analysed in the 3 planes; the sagittal, coronal and axial sections in the 3D module, and in the cross-sectional cuts in the dental volume reformatting module for detection of ERR and/or caries.
* A carious lesion will be considered present when radiolucency can be seen in enamel and/or dentine in any of the cuts.
* Caries will be graded according to severity into:

  * Incipient (less than halfway through the enamel)
  * Moderate (more than halfway through enamel but does not involve the dentino-enamel junction (DEJ)
  * Advanced (to the DEJ but does not extend more than half the distance to the pulp)
  * Severe (more than half the distance to the pulp)
* ERR will be diagnosed as clear loss of substance in the root of adjacent second molar teeth due to direct contact between it and impacted third molar.
* ERR will be graded according to severity into:

  * ERR involving less than half the dentine thickness (slight)
  * ERR involving at least half the dentine (moderate)
  * ERR involving the pulp cavity (severe)
* Severity of caries and ERR will be correlated to the study variables.
* CBCT images will be interpreted by two dental radiologists with more than 7 years experience independently; blinded from demographic data of the patients and from the results of each other.
* One of the radiologists will evaluate the images twice with a period of two weeks between the two reading sessions.
* Then inter-observational and intra-observational variability between the observers will be evaluated.

Bias:

No source of bias.

Study Size:

Based on the previous paper by Tassoker et al.1 2018, conducted in Turkey, the prevalence of ERR was 21%. Using a precision of 5, a design effect set at 1 with 95% CI (confidence interval), a total sample size of 255 will be sufficient. The sample size was calculated by Epi info.

Quantitative Variables:

The number of CBCT scans of Egyptian individuals with ERR and/or distal caries in mandibular 2nd molars associated with mandibular 3rd molars will be counted to estimate their frequency in the Egyptian population.

Statistical methods:

Data will be analysed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Comparisons between male and females for normally distributed numeric variables will be done using the Student's t-test while for non-normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be older than 18 years old.
* Having all teeth erupted except the third molar.

Exclusion Criteria:

* Completely erupted third molars.
* Impacted third molars with pathologic lesions.
* Third molars with evidence of root development which is less than two-thirds.
* Any artifact demonstration that obscure the areas of interest.
* Missing third molars.
* Patients with developmental disorders like microdontia, presence of fourth molars, impacted second molars, supernumerary teeth, and odontomes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Presence of external root resorption (ERR) in mandibular 2nd molars in percentage | Up to 2020
  Detection of external root resorption in mandibular 2nd molars associated with mandibular impacted third molars using CBCT software Romexis, (Dichotomous data - Yes/No)

SECONDARY OUTCOMES:
Presence of distal caries in mandibular 2nd molars in percentage | Up to 2020
  Detection of distal caries in mandibular 2nd molars associated with mandibular impacted third molars using CBCT software Romexis, (Dichotomous data - Yes or No )